CLINICAL TRIAL: NCT01216995
Title: A Phase II Trial of Safety and Efficacy of ADRCs Delivered Via the Intracoronary Route in the Treatment of Patients With ST-elevation Acute Myocardial Infarction - The ADVANCE Study
Brief Title: Safety and Efficacy of Adipose Derived Regenerative Cells (ADRCs) Delivered Via the Intracoronary Route in the Treatment of Patients With ST-elevation Acute Myocardial Infarction (AMI)
Acronym: ADVANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADVANCE
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Heart Attack; Regenerative Cells; Stem Cells
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose A (Active Comparator): Dose A
  Interventions: Biological: Dose A
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Dose A — ADRC Dose A
  Other Names: Adipose-Derived Regenerative Cells
  Arms: Dose A
Biological: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
Double blind, prospective, randomized, placebo-controlled Safety and Efficacy trial of ADRCs delivered via the intracoronary route in the treatment of patients with ST-elevation acute myocardial infarction (STEMI).

DETAILED DESCRIPTION:
This is a prospective, randomized, two arm, placebo-controlled, double blind, study that will enroll approximately 216 patients at no more than thirty-five (35) international clinical sites. Additional blinding measures will be taken in the assessment of study outcomes. The dose of the test material (ADRCs)is described in the protocol. The study will include two arms.

ELIGIBILITY:
Key Inclusion Criteria:

* ST-segment Elevation Myocardial Infarction (STEMI) Criteria:
* Ischemic symptoms AND
* ECG:
* Development of pathologic Q waves on the ECG; or
* ECG changes indicative of severe ischemia (ST segment elevation and/or depression); or
* New left bundle branch block; AND
* Creatine Phosphokinase Isoenzyme (MB Form) > 100 IU/L, or troponin >5x the upper limit of normal between admission and randomization
* Successful revascularization of the culprit lesion in a major epicardial vessel

Key Exclusion Criteria:

* More than 24 hours between PCI and start of liposuction
* Prior myocardial infarction, cardiomyopathy, or a history of congestive heart failure
* Pacemaker, ICD, or any other contra-indication for MRI
* Patients with increased bleeding risk
* Cardiogenic shock present post-index PCI

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction in Infarct Size | 6 Months
  Reduction in infarct size at 6 months as measured by cardiac MRI

SECONDARY OUTCOMES:
MACCE Rates | Through 36 months
  Major Adverse Cardiac and Cerebral events (MACCE) is a composite clinical endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Study Director — Cytori Therapeutics
Locations (4):
- Erasmus University Medical Centrum, Rotterdam, Netherlands
- Poland (3):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Szpital Uniwersytecki Samodzielna Pracownia Zakladu Hemodynamiki, Krakow
  - Samodzielny Publiczny Centralny Szpital Kliniczny Pracownia Kardiologii Inwazyjnej, Warsaw